CLINICAL TRIAL: NCT05732662
Title: SBRT Combined With PD-1/CTLA-4 Dual Antibody to Overcome Anti-PD-1 Resistant in Relapsed or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: SBRT Combined With AK104 to Treatment Relapsed or Metastatic ESCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Principal Investigator, Wendong Gu, chief physician, The First People's Hospital of Changzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRTAK104
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Keywords: SBRT, AK104
MeSH Terms: conditions — Recurrence; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT combined with PD-1/CTLA-4 dual antibody (Experimental)
  Interventions: Radiation: SBRT; Drug: Cadonilimab

INTERVENTIONS:
Radiation: SBRT — 24-50Gy/8-12.5Gy/3-4f
Drug: Cadonilimab — 10 mg/kg,q3w

SUMMARY:
The entire treatment process is divided into two phases: Phase I SBRT combined with PD-1/CTLA-4 bispecific antibody (AK104) and Phase II AK104 single-agent maintenance therapy.

DETAILED DESCRIPTION:
Phase I SBRT combined with AK104 treatment Target area and dose of SBRT: Select a relapsed or metastatic lymph node or lesion that has little effect on surrounding normal tissues and has not been irradiated before, and then perform radiation therapy with a total dose of 24-50Gy/8-12.5Gy/3-4f per lesion (the specific target area and dose range will be decided by the treating physician). AK104 is administered within one week after SBRT, and the regimen for AK104 is 10 mg/kg as a single dose. If multiple target lesions are treated with SBRT, multiple cycles of 21 days each are possible. When patients are treated with multiple courses of radiotherapy, it is difficult to ensure the accuracy of the overlapping doses of the re-course of radiotherapy, and the cumulative dose of organs at risk (OAR) is evaluated using the deformable image registration (DIR) technique.

Phase II AK104 monotherapy maintenance phase Monotherapy maintenance with AK104 10 mg/kg every 21 days until progression, up to one year if no progression. Patients were enrolled in Phase I and Phase II for a minimum of three cycles.

In addition, 10 mL of peripheral blood was drawn from patients before each cycle of treatment and analyzed by flow cytometry for lymphocyte subpopulation. And the changes of HMGB1 and cytokines IL-8, IL-6, IL-12, IFN-α, IFN-β, IL-2, IL-4, IL-5, INF-γ, TNF-α, IL-10, TGF-β were detected by ELISA test. By testing the above indicators, they are used to respond to the immune status after treatment as well as to screen for valid indicators that can be used to assess efficacy.

Throughout the study period, the assessment should be performed as much as possible according to the imaging assessment plan time points specified in the protocol. Tumor imaging assessments will be performed every 6 weeks during the first phase of treatment and every 9 weeks during the second phase of treatment. This project used velosity software to perform clinical tumor imaging assessment according to RECIST 1.1 criteria and irRECIST and iRECIST criteria assessment every 6 weeks; NCI-CTCAE 5.0 was used for safety assessment and adverse events were recorded throughout the study until 30 days after the end of treatment.

After the end of treatment, all subjects will be followed for survival every 3 months until death, loss to follow-up, withdrawal of knowledge, or the sponsor's decision to terminate the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. age ≥ 18 years. 2. patients enrolled must be eligible for PD-1 treatment-naïve patients with recurrent or metastatic advanced esophageal squamous carcinoma with definite measurable recurrent or metastatic lesions.

  3. have at least 2 or more clearly measurable lesions (maximum diameter of lesions≥1 cm and shortest diameter of ≥1.5 cm of lymph nodes according to RECIST v1.1), at least one of which is feasible for radiation therapy).

  4. no congestive heart failure, unstable angina, or unstable arrhythmia within the last 6 months.

  5. patient activity status score of 0-3 on the Eastern Cooperative Oncology Group (ECOG) scale with a life expectancy assessment of ≥ 3 months.

  6. no previous serious abnormalities of hematopoietic, cardiac, pulmonary, hepatic, or renal function and immunodeficiency.

  7. absolute T-lymphocyte values ≥ 0.5 times the lower limit of normal and neutrophils ≥ 2.0 × 109/L; AST and ALT ≤ 3.0 times the upper limit of normal (≤ 5.0 times the upper limit of normal for hepatocellular carcinoma/metastatic liver cancer); and creatinine ≤ 3.0 times the upper limit of normal, 1 week before enrollment.

  8. patients must have the ability to understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* 1. pregnant gestational or lactating women. 2. those with a history of other malignant diseases in the last 5 years. 3. persons with a history of uncontrolled epilepsy, central nervous system disease, or psychiatric disorder whose clinical severity, as judged by the investigator, may prevent signing an informed consent form or affect patient compliance with medication.

  4. clinically significant (i.e., active) heart disease such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or severe arrhythmias requiring pharmacologic intervention, or a history of myocardial infarction within the last 12 months.

  5. organ transplantation requiring immunosuppressive therapy. 6. Significant active infection or, in the judgment of the investigator, significant hematologic, renal, metabolic, gastrointestinal, endocrine dysfunction or metabolic disorder, or other serious uncontrolled concomitant disease.

  7. hypersensitivity to any investigational drug component. 8. have a history of immunodeficiency, including testing positive for HIV or having other acquired or congenital immunodeficiency diseases, or a history of organ transplantation, or other immune-related diseases requiring long-term oral hormone therapy.

  9. those who are undergoing acute or chronic TB infection (patients with positive T-spot test and suspicious TB foci on chest radiograph).

  10. other conditions that the investigator considers unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 3 years
  objective response rate

SECONDARY OUTCOMES:
PFS | Up to 3 years
  progression-free surviva
OS | Up to 3 years
  Overall survival
Treatment Related Severe Adverse Effects | Up to 3 years
  Number of participants with treatment-related severe adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0